CLINICAL TRIAL: NCT03654989
Title: Iontophoresis of Treprostinil to Enhance Wound Healing in Diabetic Foot Skin Ulcers
Acronym: InTREPiD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 38RC17.163
Record Dates: First submitted 2018-08-20; First posted 2018-08-31 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Diabetic Foot Ulcer
Keywords: Iontophoresis; Treprostinil; Diabetic; Foot Ulcer; Wound Healing
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer

STUDY DESIGN:
Intervention Model Description: 2 sub-studies:
  * Preliminary safety study, Phase I: single ascending dose study that aims at establishing the safety, tolerability, and PK of the procedure in patients with active ulcers; we propose an accelerated titration design with 7 doses of gel. The accelerated phase (first four doses) uses single-patient cohorts per dose. After these doses, a standard 3+3 design will be performed. Any occurrence of dose-limiting toxicity (DLT) during the accelerated phase halts the accelerated titration and the cohort is expended to the standard 3+3 design. Two instances of DLT at a dose level halt escalation, and D-1 is the maximum tolerated dose.
  * Proof-of-concept study, Phase II: Thirty-six patients with DFU associated with microvascular dysfunction will be randomized into three groups: Treprostinil iontophoresis; Placebo iontophoresis; Standard care. Drug administration, but not standard care, will be double-blind. After a 10-day treatment, follow-up includes 6 visits over 10 weeks.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Double blind (for the two groups treated with iontophoresis of treprostinil or placebo); open for the standard of care group.
  The preparation of syringes of gel containing treprostinil or placebo will be centralized. Both gels will be physically identical, and investigators will not have access to the randomization list or to preparation records. This ensures proper blinding at treatment initiation. Treatment kits will subsequently be given to research nurses to continue the treatment at home. Nurses will not have access to the randomization list or preparation records either, which guarantees proper blinding throughout the 10-day treatment.
  Unblinding will be done in case of any suspicion of an unexpected serious adverse reaction, prior to the declaration of the event to the competent authorities. Unblinding may be done 24/24h by the Pharmacy department.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Treprostinil iontophoresis (Experimental): Gel of treprostinil 1 mg/mL (target concentration)
  * Part 1: 1 administration/day, on separate days, with 72h between two doses. Ascending doses are 0.025 mg/mL, 0.05mg/mL, 0.1 mg/mL, 0.25 mg/mL, 0.5 mg/mL, 0.7 mg/mL, and 1 mg/mL. The intensity will be set at 120 µA during 60 minutes, i.e. a total current of 17.3 mC/cm².
  * Part 2: 1 administration/day at the maximum tolerated dose (MTD) for 10 days; dressing will be changed by a trained nurse every 2 days. The intensity will be set at 120 µA during 60 minutes, i.e. a total current of 17.3 mC/cm².
  Interventions: Drug: Treprostinil iontophoresis
- Remodulin® Placebo iontophoresis (Placebo Comparator): Placebo will be made from the placebo of Remodulin® incorporated into hydrogel (Suprasorb® G). The route and frequency of administration will be the same as for the investigational drug (topical administration by iontophoresis).
  Interventions: Device: Remodulin® placebo iontophoresis
- Standard care (No Intervention): subjects randomized to the standard of care group (no iontophoresis) will only undergo standard blood test at visit 0 or 1, unless tests <1 month before inclusion are available This group is not double blind Standard care consists on debridement and dressings

INTERVENTIONS:
Drug: Treprostinil iontophoresis — We will administer treprostinil at increasing doses by a iontophoresis.
  Arms: Treprostinil iontophoresis
Device: Remodulin® placebo iontophoresis — Placebo iontophoresis will be performed using Remodulin® placebo (United Therapeutics) delivered with Axion GmbH electrodes connected to a PeriIont generator (Perimed).
  * Part 1: 1 administration/day, on separate days, with 72h between two doses. The intensity will be set at 120 µA during 60 minutes, i.e. a total current of 17.3 mC/cm².
  * Part 2: 1 administration/day for 10 days. The intensity will be set at 120 µA during 60 minutes, i.e. a total current of 17.3 mC/cm².
  Arms: Remodulin® Placebo iontophoresis

SUMMARY:
Assess the effect of iontophoresis of treprostinil on wound closure over 12 weeks, in patients with DFU.

In the present study the investigators aim at establishing the proof-of-concept of iontophoresis of treprostinil as a potential treatment of diabetic foot ulcers in humans. The main hypothesis is that in patients with DFUs, the pharmacodynamic effect of a PGI2 analogue potentiates the effect of low-intensity current on microvascular function, tissue oxygenation and healing.

DETAILED DESCRIPTION:
Diabetic foot ulcers (DFUs) represent a serious public health problem associated with significant morbidity and health costs. Despite optimal etiologic treatment and local care, amputation is frequent, stressing the need for new treatments. Tissue ischemia is the primary cause for nonhealing DFUs. The cutaneous microcirculation, by providing tissue perfusion, fluid hemostasis, and delivery of oxygen and nutrients, plays a critical role in the pathophysiology and impaired healing of DFUs.

The investigators therefore hypothesize that the skin microcirculation, and more specifically the prostacyclin (PGI2) pathway, is an interesting target for the local treatment of DFUs. Indeed, besides its potent vasodilator effect, PGI2 plays a role in the promotion of fibroblast migration and angiogenesis in wound models.

However, the benefit of systemic (i.e. IV or SC) treatments is counterbalanced by potentially serious vasodilatation-induced side effects (e.g. severe headaches, flushing, tachycardia and hypotension). These properties are dose-limiting and are associated with safety issues and increased costs. The paradox is that impaired microvasculature prevents the drug, when administered intravenously, from diffusing properly to the wound. Elevated doses are therefore needed, leading to adverse drug reactions.

The originality of this approach is to locally deliver negatively charged PGI2 analogues into and around the wound under the influence of a low-intensity current, through a method called iontophoresis. Iontophoresis enables a controlled delivery of ionized drugs into/through the skin under the influence of low-intensity current. In addition, endogenous electrical signals in the wound are known to play a role in healing, by increasing the directed migration of keratinocytes, fibroblasts and neutrophils. Exogenous electric stimulation would mimic this phenomenon with a positive impact on wound healing. In summary, both the drug and its vehicle could therefore work synergistically, while delivering the drug locally therefore limiting side effects due to systemic diffusion.

This is a prospective, monocentric, controlled, randomized, double-blinded phase I/II study The main objective is to assess the effect of iontophoresis of treprostinil on wound closure over 12 weeks, in patients with DFU. The investigators will compare wound closure, expressed as the percentage change of the wound area over time (12-week follow-up), between 3 groups: iontophoresis of treprostinil, iontophoresis of placebo, and standard of care. Wound area will be assessed with a digital camera and image analysis software.

Secondary objectives are:

* To assess the effect of iontophoresis of treprostinil on complete healing over 3 months
* To assess the effect of iontophoresis of treprostinil on the time to complete healing
* To assess the effect of iontophoresis of treprostinil on skin perfusion at the site of the ulcer and around the wound
* To evaluate the effect of iontophoresis of treprostinil on skin oxygenation around the lesion and on healed skin
* To assess the pharmacokinetics (PK) of topical administration of treprostinil over damaged (wounded)
* To evaluate the safety of the procedure

The study will be divided into two consecutive parts:

Part 1: 8 to 24 patients with DFU (depending on the total number of doses tested, and the number of doses per patient) will be included in a single ascending dose (SAD) safety study of treprostinil iontophoresis.

Part 2: 36 patients with DFU associated with microvascular dysfunction (+/- neuropathy) will be randomized into three groups to receive either: 1. Treprostinil iontophoresis; 2. Placebo iontophoresis; 3. Standard care. Drug administration (placebo or treprostinil), but not standard care, will be double-blind. After a 10-day treatment, follow-up includes 6 visits over 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes according to the criteria of the American Diabetes Association (ADA), with one or more foot ulcer of microvascular or mixed etiology:

  * The ulcer size must be ≥1 cm² and <20 cm²
  * Grade 1A, 1C, 2A or 2C (University of Texas Classification of Diabetic Foot)
* Patient affiliated to social security insurance or beneficiary of social security insurance.

Exclusion Criteria:

* History of hypersensitivity reaction to treprostinil
* Pulmonary veno-occlusive disease (PVOD)
* Systemic treatment with any PGI2 analogue in the past two months.
* Critical ischemia of the lower limb, defined as leg pain at rest associated with ankle pressure <50 mmHg.
* Infected wound, treated with antibiotics in the past 15 days.
* Active or uncontrolled cardiovascular disease as follows:
* Myocardial infarction, or angina within 6 months of study participation
* Arrhythmia (uncontrolled, highly symptomatic, requires treatment or life-threatening).
* Congestive heart failure.
* Stroke or transient ischemic attack within 3 months of study participation
* Uncontrolled hypertension: systolic blood pressure> 180 mmHg or diastolic blood pressure> 105 mmHg (2 abnormal readings during visit)
* Valvular heart disease
* Severe liver disease (Child-Pugh C) at the time of enrollment
* Active gastroduodenal ulcer
* Intracerebral hemorrhage
* Trauma or any clinical event susceptible to be responsible for hemorrhage within 6 months of study participation
* Renal disease (creatinine > 2 mg/dL and/or estimated glomerular filtration rate<30 mL/min, history of dialysis)
* Unstable diabetes that has resulted in hyperosmolar coma or ketoacidosis, and/or documented increase or decrease in HbA1c of more than 2.0% within the previous 3 months.
* Pregnancy or Lactation
* Females of childbearing potential not using an effective form of birth control as determined by the investigators.
* Participant involved in another interventional clinical study
* Person deprived of liberty by judicial order
* Person under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Comparison of wound closure between the 3 groups: iontophoresis of treprostinil, iontophoresis of placebo, and standard of care, over12 weeks. | Up to 12 weeks
  Wound closure is expressed as the percentage change non-reepithelialized skin area over time (12-week follow-up), assessed with a digital camera and image analysis software.

SECONDARY OUTCOMES:
The percentage of patients with complete healing at the last follow-up visit | week 12
  Wound area will be assessed with a digital camera and image analysis software.
Comparison of time to complete healing between groups | From date of randomization until the date of documented healing, assessed up to 12 months.
  Time to complete reepithelialization will be sought in the medical record on a monthly basis.
The effect of iontophoresis of treprostinil on skin perfusion assessed with laser speckle contrast imaging at the site of the ulcer and around the wound | day 9
  Cutaneous perfusion will be assessed as cutaneous vascular conductance, and compared between groups
Comparison of skin oxygenation around the lesion and on healed skin (when possible) | Day 0 and Day 9 and week 12
  Comparison using transcutaneous pressure of oxygen
8-hour PK profile. AUC0-8 | part 1 : V1 (day0) V2 (day3 or more after V1) V3 (day3 or more after V2) V4 (day3 or more after V3), Part 2 : at days 0 and 9
  8-hour PK profile. AUC0-8 will be calculated from seven time points: immediately after the end of iontophoresis ( T0), 15 min, 30 min, 1h, 2h, 4h, and 8h
Incidence of treatment-emergent adverse events, among which hypotension, any cutaneous reaction at the site of iontophoresis, local pain, liver enzymes. | During all the study, 3 months of follow-up for every subject
  All adverse events will be rated according to the NIH Common Terminology Criteria for Adverse Events.
Evaluation of safety via blood pressure | During all the study, 3 months of following for every subject
  Blood pressure will be continuously recorded with digital photoplethysmography.
Evaluation of safety via the appearance of the wound | During all the study, 3 months of following for every subject
  Photographs of the wound will be taken and sent to investigators, blinded to the group

CONTACTS AND LOCATIONS:
Overall Officials: Cracowski Jean-luc, Professor, Principal Investigator — Clinical pharmacology unit, grenoble alpes university hospital
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided